CLINICAL TRIAL: NCT06352619
Title: Third Enhanced Control of Hypertension and Thrombectomy Stroke Domain Within A Multi-faCtorial, mulTi-arm, Multi-staGe, Randomised, gLOBal Adaptive pLatform Trial for Stroke (ACT-GLOBAL_ENCHANTED3/MT)
Brief Title: Third Enhanced Control of Hypertension and Thrombectomy Stroke Domain Within ACT-GLOBAL Adaptive Platform Trial
Acronym: ENCHANTED3/MT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: University of Calgary (Other); Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACT-GLOBAL_AIS_03
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke, Acute
Keywords: Blood Pressure; Endovascular Therapy; Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conservative SBP Control (Experimental)
  Interventions: Other: Conservative SBP Control
- Moderate SBP Control (Experimental)
  Interventions: Other: Moderate SBP Control
- Intensive SBP Control (Experimental)
  Interventions: Other: Intensive SBP Control

INTERVENTIONS:
Other: Conservative SBP Control — No or minimal treatment; if there is a need to treat a patient with a very-high (>180 mmHg) baseline SBP, then the SBP reduction is 5-10mmHg or a target is 175-180 mmHg
  Arms: Conservative SBP Control
Other: Moderate SBP Control — If the patient has a very high (>180 mmHg) or moderate high (160-180 mmHg) baseline SBP, SBP reduction is 10-20mmHg or a target of160±5 mmHg, which is higher; patients with low-high (150-160 mmHg) baseline SBP will not be treated
  Arms: Moderate SBP Control
Other: Intensive SBP Control — SBP reduction by 30-50mmHg or a target of 140±5 mmHg, which is higher
  Arms: Intensive SBP Control

SUMMARY:
Several clinical trials have produced variable conclusions regarding the effects of intensive blood pressure (BP) lowering in post-EVT acute ischaemic stroke (AIS) patients. Although two trials indicate harm from very intensive target-based treatment (SBP <130 mmHg), the others neutral effects in the SBP range 140-160 mmHg. The ENCHANTED3/MT domain of the ACT-GLOBAL platform trial aims to test different approaches to the treatment of elevated SBP in post-EVT AIS patients to find an optimal BP management strategy. ENCHANTED3/MT will randomize (1:1:1) up to 2,000 patients with SBP ≥150 mmHg post-EVT to conservative (no or minimal SBP reduction by 5-10mmHg or a target of 175-180mmHg if very-high baseline SBP [≥180mmHg]), moderate (SBP reduction by 10-20mmHg or a target of 160 ± 5, whichever is higher; no control if low-high baseline SBP [150-160mmHg]), or intensive (SBP reduction by 30-50mmHg or a target of 140±5 mmHg, whichever is higher) BP management.

DETAILED DESCRIPTION:
ACT-GLOBAL is an international, multi-factorial, multi-arm, multi-stage, randomized, adaptive platform trial designed to simultaneously evaluate multiple treatments that may improve outcomes in stroke. One domain is ENCHANTED3/MT aiming to compare three BP lowering management strategies in post-EVT AIS patients with elevated SBP determine the best approach to improve functional outcome.

Background and Rationale - Different reperfusion status may have different BP patterns. A U-shaped correlation between post-EVT BP and outcomes may exist for patients who underwent recanalisation post-EVT. In addition, different BP lowering strategy may have different safety profiles and may potentially impact differently with regards to the risk of ICH for patients with reperfusion therapy.

The controversial overall clinical effect seen in clinical trials, including ENCHANTED2/MT, OPTIMAL BP, BP TARGET, BEST II and ENCHANTED, does not resolve the question over the optimal BP control strategy following EVT. The evidence is insufficient to make sensible recommendations over the optimal BP management in this important clinical group. Thus, the Blood Pressure Domain (ENCHANTED3/MT) aims to test different treatment approaches to the control of elevated SBP post-EVT in AIS patients to find the optimal BP management that leads to improved functional status with reduced ICH and no other harms.

ENCHANTED3/MT will randomize (1:1:1) up to 2,000 patients with SBP ≥150 mmHg post-EVT to the following three BP lowering management strategies.

Primary outcome is modified Rankin scale (mRS) at 90 days analysed with utility-weighted mRS using a Bayesian hierarchical linear model. Adaptive analyses will be conducted 3-monthly with prespecified statistical triggers for superiority, inferiority and equivalence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Use of endovascular therapy (EVT) within 24 hours of symptom onset or last known well according to local guidelines;
3. Sustained high systolic blood pressure ≥150 mmHg (2 readings <10 mins apart) within 3 hours after completion of EVT.

Exclusion Criteria:

1.Any definite contraindications to BP lowering treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
modified Rankin scale | 90 days
  The mRS is a 7-outcome ordered categorical scale that assesses functional neurological status after stroke. It is not intended for use as a measure of historical functional status. It is well accepted as a standard outcome around the world in the stroke community, by patients and by regulatory authorities. The seven values and the clinical summary of the individual scores are summarized in the following:
  0 = No symptoms
  1. = No significant disability; able to carry out all usual activities
  2. = Slight disability; can look after own affairs, but unable to carry out all previous activities
  3. = Moderate disability; require some help
  4. = Moderately severe disability; unable to attend to own bodily needs without assistance
  5. = Severe disability; bedridden and requiring constant nursing care and attention
  6. = Dead

SECONDARY OUTCOMES:
Excellent functional neurological outcome | 90 days
  Excellent functional neurological outcome refers to mRS 0-1. The minimum mRS is 0 (no symptoms) while the maximum mRS is 6 (death). The higher the mRS score is the worse outcome is.
Independent functional neurological outcome | 90 days
  Independent functional neurological outcome refers to mRS 0-2. The minimum mRS is 0 (no symptoms) while the maximum mRS is 6 (death). The higher the mRS score is the worse outcome is.
Health Related Quality of Life | 90 days
  Health Related Quality of Life is based on EuroQol 5 Dimension 5 Level (EQ-5D-5L). The EQ-5D-5L is a generic instrument for describing and valuing health. It is based on a descriptive system that defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has five response categories corresponding to: no problems, slight, moderate, severe and extreme problems. The version of the instrument selected for the trial is interviewer administered either in-person, or by telemedicine or by telephone.
Mortality | 90 days
  Mortality refers to the state of being not alive.
Ordinal shift of 7 levels of modified Rankin scale | 90 days
  The modified Rankin scale (mRs) is an ordinal disability score of 7 categories (0 = no symptoms to 6 = dead). The distribution of mRs scores across its different strata in patients will be calculated.
National Institute of Health Stroke Scale (NIHSS) score | 24-48 hours
  The NIHSS is a standardized neurological examination score that is a valid and reliable measure of disability and recovery after acute stroke. Scores range from 0 to 42, with higher scores indicating increasing severity. The scale includes measures of level of consciousness, extra ocular movements, motor and sensory tests, coordination, language, and speech evaluations. The NIHSS will be administered at Baseline prior to each domain randomisation (unless specified otherwise in specific domains) and Day 2. The NIHSS as part of standard of care treatment may be used if an assessment was not done by clinical trial personnel.
Any intracranial haemorrhage (ICH) | 2 days
  Any ICH is defined as ICH of any type on brain imaging ≤2 days of treatment, identified by adjudicators.
Symptomatic intracerebral haemorrhage (sICH) | 2 days
  Symptomatic ICH on follow-up imaging (up to 2 days from randomization) will be a reportable serious adverse event that is adjudicated centrally according to the standard approach of reporting symptomatic ICHs used in the Heidelberg classification.
Serious Adverse Event (SAE) | 4 days
  As defined by the WHO International Drug Monitoring Centre (1994), an SAE is any untoward medical occurrence that is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; be an important medical event that may not result in death, be life-threatening, or require hospitalization, but may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes previously listed.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, PhD, Principal Investigator — The George Institute
Locations (2):
- The George Institute for Global Health, Sydney, New South Wales, Australia
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
After this domain is completed, the archived de-identified limited dataset of randomized participants will be transmitted to and stored in the ACT-GLOBAL Data Repository, for use by researchers. Data can be shared after publication of the main results.
Supporting Information: Study Protocol
Time Frame: Data can be shared after publication of the main results.
Access Criteria: Data can be shared after publication of the main results, based on approval of a submitted protocol to the Publication Committee. Data can be shared to bona fide researchers with experience in medical research, and with no conflict of interest that may potentially influence their interpretation of any analyses, and employed by a recognised academic institute, health service organisation, commercial research organisation of from the pharmaceutical industry. The data sharing will be only for analyses within the constraints of the consent under which the data were originally gathered consent.
  Data sharing with industry will be according to relevant contracts with appropriate approvals from all stake holders.

REFERENCES:
- See also: ACT-GLOBAL Master Protocol Registration — https://clinicaltrials.gov/study/NCT06352632